CLINICAL TRIAL: NCT01062477
Title: Safety and Immunogenicity of the Sanofi Pasteur's DTaP//PRP-T Combined Vaccine (ACTACEL) Versus Local DTaP and Hib Conjugate (Act-HIB) Monovalent Vaccine as a Three-dose Primary and Booster Vaccination in Healthy Infants in China
Brief Title: A Study of DTaP//PRP-T Combined Vaccine (ACTACEL) Versus Local DTaP and Act-HIB Monovalent Vaccine in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C5A06; UTN: U1111-1112-2509 (Other: WHO)
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Diphtheria; Tetanus; Pertussis; Haemophilus Influenzae Type B
Keywords: Diphtheria Tetanus Pertussis Haemophilus Influenzae Type B
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Haemophilus Infections | interventions — Hiberix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Study Group 1 (Experimental): Participants will receive ACTACEL vaccine at 2, 3, and 4 months of age.
  Interventions: Biological: DTaP//PRP-T Combined Vaccine
- Study Group 2 (Experimental): Participants will receive ACTACEL vaccine at 3, 4, and 5 months of age.
  Interventions: Biological: DTaP//PRP-T Combined Vaccine
- Study Group 3 (Active Comparator): Participants will receive Wuhan DTaP and Act-HIB vaccines concomitantly at 3, 4 and 5 months of age.
  Interventions: Biological: DTaP Combined Vaccine and PRP-Tetanus Conjugate Vaccine

INTERVENTIONS:
Biological: DTaP//PRP-T Combined Vaccine — 0.5 mL, Intramuscular
  Other Names: ACTACEL
  Arms: Study Group 1
Biological: DTaP//PRP-T Combined Vaccine — 0.5 mL, Intramuscular
  Other Names: ACTACEL
  Arms: Study Group 2
Biological: DTaP Combined Vaccine and PRP-Tetanus Conjugate Vaccine — 0.5 mL, Intramuscular (each vaccine)
  Other Names: Act-HIB™
  Arms: Study Group 3

SUMMARY:
The purpose of this study is to assess the immunogenicity and safety of ACTACEL combined vaccine in support of registration of this product in China

Primary Objectives:

* To demonstrate that ACTACEL vaccine administered at 2, 3 and 4 months of age or at 3, 4 and 5 months of age is not inferior, in terms of seroprotection, to Wuhan's Diphtheria, Tetanus, acellular Pertussis (DTaP) and Haemophilus influenzae type b (Act-HIB) vaccine given concomitantly, for diphtheria, tetanus, and Polyribosyl Ribitol Phosphate (PRP) antigens, one month after the three-dose primary vaccination.
* To demonstrate the superiority, in terms of seroconversion, of ACTACEL vaccine administered at 2, 3 and 4 months of age or at 3, 4 and 5 months of age for Pertussis Toxoid (PT), Fimbriae types 2 and 3 (FIM2) and (FIM3) pertussis antigens, compared with Wuhan's DTaP and Act-HIB vaccines given concomitantly, one month after the three-dose primary vaccination.

Secondary Objectives:

* To describe the safety after administration of the study vaccines.
* To describe in each group the immunogenicity of the study vaccines one month after the primary vaccination and before and one month after the booster vaccination.

DETAILED DESCRIPTION:
Participants will receive a primary vaccination consisting of three doses of ACTACEL at either 2, 3, and 4 months of age or at 3, 4, and 5 months of age; or Wuhan DTaP and Act-HIB vaccines at 3, 4, and 5 months of age. All participants will receive a single booster dose at 18-20 months of age and will be followed up for one month after the last dose of study vaccine.

ELIGIBILITY:
Inclusion Criteria :

* Aged 2 months on the day of inclusion
* Born at full term pregnancy (≥ 36 weeks) with a birth weight ≥ 2.5 kg
* Informed consent form signed by the parent(s) or legal representative
* Participant and parent/legal representative able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria :

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy since birth, or long-term systemic corticosteroids therapy
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator
* Receipt of blood or blood-derived products since birth that might interfere with the assessment of immune response
* Receipt or planned receipt of any vaccine in the 4 weeks preceding or following any trial vaccination (except oral poliovirus (OPV), bacillus Calmette-Guérin (BCG), and Hepatitis B vaccines which cannot be given within 8 days before or after any study vaccination)
* History of seizures
* Known personal or maternal Human Immunodeficiency Virus (HIV), Hepatitis B (HB) surface antigen or Hepatitis C seropositivity
* History of diphtheria, tetanus, pertussis or Haemophilus influenzae type b infection (confirmed either clinically, serologically or microbiologically)
* Previous vaccination against diphtheria, tetanus, pertussis or Haemophilus influenzae type b disease with either the trial vaccine or another vaccine
* Participant at high risk for diphtheria, tetanus, pertussis or Haemophilus influenzae type b infection during the trial
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular vaccination
* History of contraindication to vaccination with pertussis-containing vaccine
* Febrile illness (axillary temperature ≥37.1°C) or moderate or severe acute illness/infection on the day of inclusion, according to Investigator judgment

Temporary contraindications that must be resolved before vaccination:

* Acute febrile illness within the 72 hours preceding the vaccination, or temperature ≥37.1°C present at this visit
* Any vaccination in the 4 weeks preceding the vaccination (except OPV, BCG, and hepatitis B vaccines which cannot be given within 8 days before or after any study vaccination)
* Systemic corticosteroids therapy (prednisone or equivalent) for more than 2 consecutive weeks within the past 3 months

Ages: 60 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1056 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: To provide information concerning the immunogenicity of ACTACEL vaccine after primary and booster vaccination. | One month post-vaccination

SECONDARY OUTCOMES:
Safety: To provide information concerning the safety after primary and booster administration of ACTACEL vaccine. | 0-7 days post-vaccination and entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- China (2):
  - LingChuan County, Guilin City, Guangxi
  - Lipu County, Guilin City, Guangxi

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com